CLINICAL TRIAL: NCT00196274
Title: Autonomic Regulation Trial (ART)
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Other Study IDs: GE IDE No. R00500; BMBF13N7705/2
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2005-09

CONDITIONS: Infarction, Myocardial
Keywords: AUTONOMIC NERVOUS SYSTEM; Assessment, Risk
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study was to develope and evaluate a new method for risk stratification which predicts high mortality risk in patients with cardiac disease based on simultateous examination of high resolution ECG, continuous arterial pressure and a breathing signal.

ELIGIBILITY:
Inclusion Criteria:

acute myocardial infarction, presence of sinus rhythm

Exclusion Criteria:

diseases (other than acute myocardial infarction) with impact on prognosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmidt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Petra Barthel, MD, Study Director — Deutsches Herzzentrum Muenchen; Axel Bauer, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Schmidt G, Malik M, Barthel P, Schneider R, Ulm K, Rolnitzky L, Camm AJ, Bigger JT Jr, Schomig A. Heart-rate turbulence after ventricular premature beats as a predictor of mortality after acute myocardial infarction. Lancet. 1999 Apr 24;353(9162):1390-6. doi: 10.1016/S0140-6736(98)08428-1. PMID 10227219
- [Background] Barthel P, Schneider R, Bauer A, Ulm K, Schmitt C, Schomig A, Schmidt G. Risk stratification after acute myocardial infarction by heart rate turbulence. Circulation. 2003 Sep 9;108(10):1221-6. doi: 10.1161/01.CIR.0000088783.34082.89. Epub 2003 Aug 25. PMID 12939209
- [Background] Makikallio TH, Barthel P, Schneider R, Bauer A, Tapanainen JM, Tulppo MP, Schmidt G, Huikuri HV. Prediction of sudden cardiac death after acute myocardial infarction: role of Holter monitoring in the modern treatment era. Eur Heart J. 2005 Apr;26(8):762-9. doi: 10.1093/eurheartj/ehi188. Epub 2005 Mar 18. PMID 15778204
- [Background] Bauer A, Guzik P, Barthel P, Schneider R, Ulm K, Watanabe MA, Schmidt G. Reduced prognostic power of ventricular late potentials in post-infarction patients of the reperfusion era. Eur Heart J. 2005 Apr;26(8):755-61. doi: 10.1093/eurheartj/ehi101. Epub 2005 Jan 26. PMID 15673543
- [Derived] El-Hamad FJ, Bonabi SY, Muller A, Steger A, Schmidt G, Baumert M. Augmented Oscillations in QT Interval Duration Predict Mortality Post Myocardial Infarction Independent of Heart Rate. Front Physiol. 2020 Nov 9;11:578173. doi: 10.3389/fphys.2020.578173. eCollection 2020. PMID 33240101
- [Derived] Sinnecker D, Dirschinger RJ, Barthel P, Muller A, Morley-Davies A, Hapfelmeier A, Dommasch M, Huster KM, Hasenfuss G, Laugwitz KL, Malik M, Schmidt G. Postextrasystolic blood pressure potentiation predicts poor outcome of cardiac patients. J Am Heart Assoc. 2014 Jun 3;3(3):e000857. doi: 10.1161/JAHA.114.000857. PMID 24895163
- [Derived] Rizas KD, Nieminen T, Barthel P, Zurn CS, Kahonen M, Viik J, Lehtimaki T, Nikus K, Eick C, Greiner TO, Wendel HP, Seizer P, Schreieck J, Gawaz M, Schmidt G, Bauer A. Sympathetic activity-associated periodic repolarization dynamics predict mortality following myocardial infarction. J Clin Invest. 2014 Apr;124(4):1770-80. doi: 10.1172/JCI70085. Epub 2014 Mar 18. PMID 24642467